CLINICAL TRIAL: NCT04906863
Title: Genetic Studies of Early-onset Dementia
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: University of Miami (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Christiane Reitz, MD, PhD, Associate Professor of Neurology and Epidemiology, Columbia University
Other Study IDs: AAAQ9793; 5U24AG056270-07 (NIH); 1R01AG064614 (NIH)
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Dementia, Early Onset
Keywords: Alzheimer's Disease; Memory loss; Early-onset Alzheimer's disease; Mild cognitive impairment; Normal cognition; Dementia; Genetics
MeSH Terms: conditions — Dementia; Alzheimer Disease; Memory Disorders; Cognitive Dysfunction | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 40ml of blood and/or saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild Cognitive Impairment: Individuals with mild cognitive impairment that began before age 70
  Interventions: Genetic: Blood draw; Other: Neurocognitive testing; Other: Medical questionnaire
- Dementia/Alzheimer's Disease: Individuals with Alzheimer's Disease or other dementia that began before age 70
  Interventions: Genetic: Blood draw; Other: Neurocognitive testing; Other: Medical questionnaire
- Cognitively Healthy: Cognitively healthy individuals over the age of 30 years
  Interventions: Genetic: Blood draw; Other: Neurocognitive testing; Other: Medical questionnaire

INTERVENTIONS:
Genetic: Blood draw — Blood draw for identification of genetic variants associated with the development of memory problems
Other: Neurocognitive testing — Brief memory test
Other: Medical questionnaire — Collection of medical history

SUMMARY:
The aim of this study is to identify genetic factors that contribute to risk and progression of early-onset dementia (loss of memory function before the age of 70 years) across all ethnic groups, including Alzheimer's Disease, mild cognitive impairment and other dementias.

DETAILED DESCRIPTION:
The study population includes individuals affected by Alzheimer's Disease, mild cognitive impairment, other dementias, cognitively healthy individuals without memory problems, or their family members.

Ascertainment is across both males and females, and all race and ethnic groups.

ELIGIBILITY:
Inclusion criteria:

* 18 years and older
* Individuals diagnosed with dementia, their family members and unrelated healthy controls without dementia.

Exclusion Criteria:

-Individuals with competing diagnosis such as Huntington's disease, traumatic brain injury, drug or alcohol abuse, or schizophrenia, etc., unless family members of a dementia affected individual

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals affected by dementia, mild cognitive impairment, cognitively healthy individuals, or their family members. Ascertainment is across both males and females, and all race-ethnic groups.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-09-14 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Genetic risk variants associated with early-onset dementia | 2 years
  Genetic factors will be measured through genome-wide genotyping arrays and/or whole-genome sequencing, and then correlated with Alzheimer disease and related phenotypes, such as cognitive impairment, functional impairment, and relevant biomarkers.
Changes in blood biomarkers in early-onset dementia | 2 years
  Blood biomarkers including plasma amyloid beta and tau protein will be assessed in blood and correlated with onset and progression of memory loss and functional impairment

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Reitz, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be shared via government required repositories and with our collaborators. Data are coded, with no personally identifiable information included. Data shared include the genomic data (array data, sequence data, APOE genotyping results, etc), phenotype data (case/control status, age of onset, etc), and basic demographic information (sex, race/ethnicity data if available, etc).
  The NIH Genomic Data Sharing Policy (GDS Policy) took effect on January 25th, 2015. This necessitates that we send coded data and samples to the National Institute on Aging Genetics of Alzheimer's Disease (NIAGADS)l; in some cases materials derived from participants (blood or DNA) may be stored at the National Cell Repository for Alzheimer's Disease (NCRAD).
  We may share deidentified genomic and phenotypic data with collaborators at other sites in order the accomplish the scientific aims of the study. Such research is performed with the approval of the local internal review boards.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: This study adheres to the NIA Alzheimer Disease Genomics Data Sharing Plan (https://www.nia.nih.gov/research/dn/alzheimers-disease-genomics-sharing-plan). As such, genomic data will be deposited in NIH/NIA data repositories (www.niagads.org). For genomic data, this typically happens within a year of data generation, or upon publication in scientific journals (whichever is sooner). Basic phenotypic data (affection status, age of onset, sex, family structure if applicable, etc) are deposited with the genomic data. More detailed phenotypic data (cognitive data, biomarker, etc) will be made available upon publication. Data dictionaries for primary data (genomic data and basic phenotypic data) will be available with the deposition of data into the NIH/NIA data repositories (www.niagads.org). Additional supporting documentation (analysis plans, study protocols, etc) is typically described in detail upon publication of results in peer reviewed literature.
Access Criteria: This study adheres to the NIA Alzheimer disease Genomics Data Sharing Plan (https://www.nia.nih.gov/research/dn/alzheimers-disease-genomics-sharing-plan). As part of this plan data distribution agreements are required before recipients receive any data from this study. The primary requirements for the DDA include language ensuring that (1) data are not transferred to others beyond the initial recipient, (2) no attempt will be made to identify participants, (3) any results or data generated as part of the study will be shared back to NIA/NIAGADS. See the NIA Data Distribution Agreement for more details (https://www.niagads.org/sites/all/public_files/NIAGADS-DDA.pdf).
URL: https://www.nia.nih.gov/research/dn/alzheimers-disease-genomics-sharing-plan